CLINICAL TRIAL: NCT06373315
Title: The Effect of Smartphone and Hand Anthropometry on Pain and Upper Extremity Functions
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Feyza Altindal Karabulut, Assistant Professor, Nigde Omer Halisdemir University
Other Study IDs: 2023/11-18
Record Dates: First submitted 2024-04-02; First posted 2024-04-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Upper Extremity Problem; Smartphone Addiction
Keywords: Anthropometric Measurements; Upper Extremity; Smartphone
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sample of Study: Volunteer participants who constitute the study sample include students and staff studying in different departments at the university. Inclusion criteria; It includes using a smartphone for more than 1 hour a day to send at least 5 emails or text messages a day, play games or browse the internet. Exclusion criteria; It includes students who have an existing injury to the hand or upper extremity (6 months ago) and who have been diagnosed with degenerative, inflammatory, musculoskeletal, neuromuscular and congenital disorders of the hand or upper extremity that affect their use in daily life.

SUMMARY:
Mobile phones have different uses in different disciplines, and this encourages long-term use. For optimum comfort use, it is important to ensure users' awareness when purchasing mobile phones that match their hand sizes. The number of studies in the literature on this subject is limited. In this context, the aim of our study is to investigate the relationship between smartphone and hand anthropometry measurements and upper extremity pain and functions.

DETAILED DESCRIPTION:
Phone design features cause different problems on body mechanics and musculoskeletal system. With the use of smartphones, people tend to maintain incorrect postures for long periods of time, which increases tension in the body. This situation causes complaints such as cervical disc herniation, tingling complaints in different body parts, overuse injuries, Upper Crosses syndrome, and carpal tunnel syndrome. On the other hand, the use of smartphones is increasing among students for reasons such as providing students with freedom of time and space, increasing the speed of teaching and learning, supporting one-on-one learning, and increasing the number of ideas produced by encouraging a group discussion environment.

Mobile phones have different uses in different disciplines, and this encourages long-term use. Although many musculoskeletal system structures can be affected by incorrect postures due to the long-term use of smart mobile phones, it is thought that the upper extremity is most affected. Therefore, the aim of our study is to investigate the relationship between smartphone dimensions and hand anthropometric measurements and upper extremity pain and functions in order to raise awareness when purchasing mobile phones that match users' hand sizes for optimum comfort and use.

ELIGIBILITY:
Inclusion Criteria:

* Sending at least 5 e-mails or text messages a day from your mobile phone,
* Using a smartphone for more than 1 hour a day to play games or browse the internet

Exclusion Criteria:

* Having an existing injury in the hand or upper extremity (suffered 6 months ago)
* Having been diagnosed with a degenerative, inflammatory, musculoskeletal, neuromuscular, or congenital disorder of the hand or upper extremity.

Ages: 17 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Volunteer participants include students and staff studying in different departments at the university.
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Hand anthropometric measurements: Hand length | 2 month
  It is the longitudinal distance in centimeters from the midpoint of the distance from the most distal styloid process of the radius to the most distal styloid process of the ulna to the tip of the 3rd finger. Measurements will be made with the participants sitting on a chair, with their hands held on a horizontal platform. While the fingers are kept as close to each other as possible in all measurements, participants will be asked to open their hands as much as they can only in the maximum hand spread measurement.
Hand anthropometric measurements: Palm length | 2 month
  It is the longitudinal distance in centimeters between the midpoint of the wrist crease and the highest point of the 3rd Metacarpal head. Measurements will be made with the participants sitting on a chair, with their hands held on a horizontal platform. While the fingers are kept as close to each other as possible in all measurements, participants will be asked to open their hands as much as they can only in the maximum hand spread measurement.
Hand anthropometric measurements: Width of the hand (Metacarpal) | 2 month
  It is the longitudinal distance in centimeters between the base of the 2nd Metacarpal bone and the base of the 5th Metacarpal bone. Measurements will be made with the participants sitting on a chair, with their hands held on a horizontal platform. While the fingers are kept as close to each other as possible in all measurements, participants will be asked to open their hands as much as they can only in the maximum hand spread measurement.
Hand anthropometric measurements: Maximum hand spread measurement | 2 month
  It is the longest distance in centimeters from the thumb to the tip of the 5th finger when your hand is open. Measurements will be made with the participants sitting on a chair, with their hands held on a horizontal platform. While the fingers are kept as close to each other as possible in all measurements, participants will be asked to open their hands as much as they can only in the maximum hand spread measurement.
Gross grip strength measurement | 2 month
  Grip strength will be measured in Newton using a Hydraulic Hand Dynamometer. Standard grip strength testing position recommended by the American Society of Hand Therapists (ASHT); Participants will sit upright on the back of a chair without armrests with their feet flat on the floor, shoulder in adduction and neutral rotation, elbow in 90 degree flexion, forearm in neutral, wrist in slight extension and (0-150) degree ulnar deviation. It will be measured 3 times, and a 1-minute rest break will be given between each trial. The average of 3 attempts will be calculated for each hand.
Pinch grip strength | 2 month
  Measurement of pinch grip strength in Newton will be performed with a digital pinchmeter. Pinch grip strength test position recommended by the American Society of Hand Therapists (ASHT); Participants will sit upright on the back of a chair without armrests with their feet flat on the floor, shoulder adduction and neutral rotation, elbow 90 degree flexion, forearm neutral, wrist slightly extended and (0-150) degree ulnar deviation. It will be measured 3 times, and a 1-minute rest break will be given between each trial. The average of 3 attempts will be calculated for each hand.
Measurement of phone dimensions | 2 month
  The size of the touch screen will be measured in inches diagonally from one corner of the screen to the opposite corner (6). iPhone 5 models from Apple and 6 models from Samsung Galaxy, Realme, Xiaomi Redmi, Oppo, Huawei, Infinix, Reeder and other touch screen phones will be used. Screen dimensions will be measured using a standard ruler 30 cm diagonally across the screen (3). According to screen size, mobile phones will be grouped into small, medium and large phone sizes as shown in Table 2.
Upper extremity functional status assessment | 2 month
  Quick-DASH is an evaluation questionnaire that measures activity and participation limitations in all upper extremity disorders. In the survey, patients' difficulties during daily living activities are questioned with 11 questions. Each answer is scored on a Likert scale from 1 to 5, from best to worst. There are also optionally completed Business Model (DASH-W) sections consisting of 4 questions and Sports and Musicians Model (DASH-SM) sections consisting of 4 questions. The validity and reliability of this questionnaire in Turkish was determined by Düger et al. made by. The total score for the first section consisting of 30 questions varies between 0 and 100. The total score for the second part ranges from 0 to 100. For the third part, which evaluates high performance sports, the total score varies between 0 and 100. An increase in the score in the survey indicates a decrease in functionality.

SECONDARY OUTCOMES:
Pain assessment | 2 month
  Visual Analog Scale (VAS) Standard 10 centimeters VAS (0 = "no pain", 10 = "unbearable pain") was used to determine the pain levels of the volunteers participating in the study.
Smartphone addiction | 2 month
  In our study, the Smartphone Addiction Scale Short Form, whose Turkish adaptation is valid and reliable, will be used to measure the smartphone addiction of the participants. The total number of items of this single-factor scale is 10. The scale is evaluated with a six-point Likert-type scale, and each item is scored from one (strongly disagree) to six (strongly agree). The lowest score that can be obtained from this scale is 10 and the highest score is 60. The cut-off value for the scale was found to be 31 points for men and 33 points for women. High scores from the scale indicate an increased risk of smartphone addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Altindal Karabulut, Asst. Prof., Principal Investigator — Niğde Ömer Halisdemir University; Nihal BUKER, Prof., Study Chair — Pamukkale University
Locations (1):
- Nigde Omer Halisdemir University, Bor Faculty of Health Sciences, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kamel DM, Hakeem CA, Tantawy SA. Influence of hand and smartphone anthropometric measurements on hand pain and discomfort: A cross-sectional study. Medicine (Baltimore). 2020 Mar;99(11):e19513. doi: 10.1097/MD.0000000000019513. PMID 32176099
- [Background] Werle S, Goldhahn J, Drerup S, Simmen BR, Sprott H, Herren DB. Age- and gender-specific normative data of grip and pinch strength in a healthy adult Swiss population. J Hand Surg Eur Vol. 2009 Feb;34(1):76-84. doi: 10.1177/1753193408096763. Epub 2009 Jan 7. PMID 19129352